CLINICAL TRIAL: NCT05908344
Title: Use of the Frequen-ZZZ Sleep Pad to Increase Restorative Sleep: A Proof-of-Concept Study
Brief Title: Frequen-ZZZ SleepPad Investigational Device POC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kunasan Inc. (Industry)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: Kunasan
Record Dates: First submitted 2023-06-01; First posted 2023-06-18 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-05

CONDITIONS: Insomnia; Sleep; Sleep Disturbance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Intervention Model Description: All participants in this study will experience all study conditions (i.e. a sham (Control) and an active (Intervention) Sleep Pad bedside controller device) in a randomized crossover design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is a double-blind trial, in which bedside controllers for Sleep Pad systems are coded and either "activated" or "deactivated" (sham/control) by the manufacturer prior to receipt for use in the research. A "deactivated" Sleep Pad bedside controller retains all functionality (and evidence of functionality) of an "activated" bedside controller Sleep Pad, excepting the stimulation. The blind is maintained by a designated study team member who will have access to the list linking device code IDs to their relative active/sham group, and who does not have interaction with study participants. This blind will be lifted if relevant for safety reasons in cases of serious adverse event on a participant case-by-case basis, and on the whole for other researchers after completion of the entire trial for interpretation of analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Activated Sleep Pad controller (Experimental): Treatment dosing is under participant control, by physical proximity/orientation to the Sleep Pad pad portion of the Sleep Pad system, and by a manually operated power button on an activated bedside controller portion of the Sleep Pad system. Dosing is pre-set at a stable level across all participants. Dosing occurs throughout a participant's typical nocturnal sleep period, nightly, unless manually paused by the participant.
  Interventions: Device: Activated Sleep Pad system (Frequen-ZZZ)
- Deactivated Sleep Pad controller (Sham Comparator): Use of the Sleep Pad system is consistent with the Experimental arm, excepting that a deactivated bedside controller portion of the Sleep Pad system is used.
  Interventions: Device: Deactivated Sleep Pad system (Frequen-ZZZ)

INTERVENTIONS:
Device: Activated Sleep Pad system (Frequen-ZZZ) — The investigational device is a sleep pad and bedside controller system capable of producing a low-level radio-frequency field potential. An individual laying in the correct orientation and with correct contact distance from the pad portion of a powered device experiences its specific area of effect. The field potentials generated by the pad are hypothesized to have benefit for sleep.
  Arms: Activated Sleep Pad controller
Device: Deactivated Sleep Pad system (Frequen-ZZZ) — The investigational device is a sleep pad and bedside controller system that produces a low-level radio-frequency field potential. An individual laying in the correct orientation and with correct contact distance from the pad portion of a non-powered device experiences all functional aspects of the device except the intended magnetic field potential that is hypothesized to have benefit for sleep.
  Arms: Deactivated Sleep Pad controller

SUMMARY:
The investigators propose to examine the potential effects of the Frequen- ZZZ sleep pad - a noninvasive, unobtrusive appliance that generates a localized low-level electromagnetic field via radiofrequency, and that is used on the bed - on multiple sleep outcomes in an 8-week randomized crossover study, and to calculate the effect sizes of the intervention to inform power and sample size for future studies.

DETAILED DESCRIPTION:
This research is a small, 8wk clinical trial testing the potential effects of an investigational device, Frequen-ZZZ Sleep Pad, on the sleep of adults 40-65 years old. The investigators aim to determine whether sleeping with the Sleep Pad, which creates a radio-frequency field around the sleeper, improves sleep. Sleep will be primarily measured using a noninvasive clinical standard method, called polysomnography (PSG), for 6 separate nights in the personal residence of participants. Sleep will also be measured both day and night with a watch-like device that measures activity, and with surveys. The investigators will look for changes in sleep quality, in sleep duration, and in the way that sleep is organized by the body ("sleep architecture"). There are 12-15 in-person appointments across the course of the study. With the data, the investigators hope to also evaluate the feasibility and effect sizes of this non-pharmacological intervention to inform future research, and plan to use data in support of a future FDA application for the device.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is obtained from the subject.
2. Subject is an English speaker and reader. They are able to understand the procedures related to the study.
3. Subject is 40-65 years of age at enrollment (by self report at Screening & verified with photo ID at full Consent)
4. Subject is not engaged in rotating or nocturnal shift employment (by self-report at Screening)
5. Subject is living independently (by self-report and/or according to their status at a community living facility)
6. Subject's personal residence is equipped with functional WiFi and subject is willing to permit study device connection to their WiFi (by self-report at Screening)
7. Insomnia Severity Index score of ≥8 at enrollment (based on self-administration at screening)
8. Willing to refrain from initiating new, sleep-directed interventions (e.g. medication; behavioral) that are not a part of this study protocol for the duration of study participation (by self-report)
9. Willing to refrain from all nicotine use for the duration of participation (by self-report)
10. Willing to refrain from pet access to the bed or sleeping space for the duration of participation (by self-report)
11. Regularly sleeping on a non-water bed (by self-report)
12. Has and uses own smart phone or tablet device, and is willing to continue to use personal device daily for study purposes (by self-report)

Exclusion Criteria:

1. Diagnosed with a sleep disorder (by self-report)
2. Has an implanted medical device (e.g., pacemaker, cochlear; by self-report)
3. Diagnosed serious mental/neurologic health disorder or substance use disorder (e.g., autism, psychosis, depression/bipolar, dementia; by self-report)
4. Personal health history of epilepsy or traumatic brain injury (by self-report)
5. Taking any physician-directed pharmacologic intervention for sleep or actively engaged in a clinically-validated course of therapy (including behavioral therapy for sleep; by self-report)
6. Diagnosed hydration problems or taking prescribed diuretic medication (by self-report)
7. Pregnant, breast-feeding, or planning to become pregnant during the study participation period (by self-report)
8. History of negative reaction to acupuncture (by self-report)
9. Recreational use of illicit substances in the past month (by self-report)
10. Any nicotine use in the past 3 months (by self-report)
11. History of sensitivity to, or considers oneself to be uniquely sensitive to, radio-frequency (by self-report)
12. Was previously engaged in this research as a randomized participant
13. If a participant does not live within a reasonable commutable distance from the Penn State University - University Park campus (i.e. ~20min) to accommodate off-site study visits, then they must be willing to accept the costs and responsibilities of coming to campus (15-17 visits) in order to participate

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Convenience sample of 40-65y/o with evidence of Insomnia symptoms in the State College, PA region.
Pre-assignment Details: Demonstrated adherence to study procedures (surveys & actigraphy worn) during Baseline (Wk 1)
Groups:
- Active Device in Phase 1, Then Sham Device in Phase 2: Wks 2-5 Active Device, Wks 6-8 Sham Device
- Sham Device in Phase 1, Then Active Device in Phase 2: Wks 2-5 Sham Device, Wks 6-8 Active Device
Period: Overall Study
Arm/Group | Active Device in Phase 1, Then Sham Device in Phase 2 | Sham Device in Phase 1, Then Active Device in Phase 2
Started | 5 | 5
Started Phase 1 | 5 | 5
Started Phase 2 | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Device Phase 1, Then Sham Device Phase 2: Wks 2-5 Active Device, then Wks 6-8 Sham Device
- Sham Device Phase 1, Then Active Device Phase 2: Wks 2-5 Sham Device, then Wks 6-8 Active Device
- Total: Total of all reporting groups
Arm/Group | Active Device Phase 1, Then Sham Device Phase 2 | Sham Device Phase 1, Then Active Device Phase 2 | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.4 (3.2) | 55.1 (8.5) | 55.2 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: Overall sum score] — Self-reported score on the Insomnia Severity Index (ISI; 0-28) e-survey, where a higher score indicates worse/more Insomnia symptoms.
  Overall sum score | 9.6 (5.2) | 12.4 (3.3) | 11.0 (4.3)
Non-Rapid Eye Movement Stage 1 (NREM1) minutes [Mean (Standard Deviation); unit: Minutes] | 61.6 (16.1) | 92.3 (61.9) | 77.0 (45.6)
Non-Rapid Eye Movement Stage 1 (NREM1) percentage [Mean (Standard Deviation); unit: % of Total Sleep] | 17.0 (5.8) | 21.7 (13.3) | 19.4 (10.0)
Non-Rapid Eye Movement Stage 2 (NREM2) minutes [Mean (Standard Deviation); unit: Minutes] | 190.2 (56.2) | 193.5 (20.9) | 191.9 (40.0)
Non-Rapid Eye Movement Stage 2 (NREM2) percentage [Mean (Standard Deviation); unit: % of Total Sleep] | 49.9 (8.5) | 47.4 (8.3) | 48.7 (8.1)
Non-Rapid Eye Movement Stage 3 (NREM3) minutes [Mean (Standard Deviation); unit: Minutes] | 20.2 (22.2) | 29.1 (30.9) | 24.7 (25.8)
Non-Rapid Eye Movement Stage 3 (NREM3) percentage [Mean (Standard Deviation); unit: % of Total Sleep] | 5.2 (5.4) | 7.2 (7.5) | 6.21 (6.26)
Rapid Eye Movement (REM) minutes [Mean (Standard Deviation); unit: Minutes] | 102.9 (17.6) | 98.0 (23.2) | 100.5 (19.6)
Rapid Eye Movement (REM) percentage [Mean (Standard Deviation); unit: % of Total Sleep] | 27.9 (6.0) | 23.7 (4.7) | 25.8 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sleep Architecture
Description: Quantity of each sleep stage defined by the American Academy of Sleep Medicine (NREM1, NREM2, NREM3, and REM), measured by clinically standard elements of Polysomnography and scored by a Registered Polysomnographic Technologist.
  Note: Randomization to Active or Sham during Phase 1 or Phase 2 occurred at the end of Baseline week.
Time Frame: The later viable night of two recordings: At the end of Phase 1 - Week 2 or Phase 1 - Week 3, and At the end of Phase 2 - Week 2 or Phase 2 - Week 3. Sleep stage minutes (relative to Latency to Persistent Sleep, Edinger et al. 2013).
Population: The same 10 (total) participants are represented in Arm/Group (repeated-measures).
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Active Device: 3wks (either study wks 2-4 in an 'Active' Phase 1 or wks 6-8 in an 'Active' Phase 2), Active bedside controller.
- Sham Device: 3wks (either study wks 2-4 in a 'Sham' Phase 1 or wks 6-8 in a 'Sham' Phase 2), Sham bedside controller.
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 10 | 10
Minutes
  NREM1 | 48.8 (23.5) | 54.0 (36.4)
  NREM2 | 212.5 (37.8) | 218.7 (40.5)
  NREM3 | 32.85 (25.8) | 22.85 (17.0)
  REM | 88.5 (32.7) | 108.9 (38.6)
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Comparison for NREM1 minutes. Group Selection refers to study device Condition (Active/Sham); repeated-measures design; Test type: Other — Effect size determination; Cohen's d = -0.24
Statistical Analysis 2: Comparison: Active Device vs Sham Device; Comparison for NREM2 minutes. Group Selection refers to study device Condition (Active/Sham); repeated-measures design; Test type: Other — Effect size determination; Cohen's d = -0.15
Statistical Analysis 3: Comparison: Active Device vs Sham Device; Comparison for NREM3 minutes. Group Selection refers to study device Condition (Active/Sham); repeated-measures design; Test type: Other — Effect size determination; Cohen's d = 0.69
Statistical Analysis 4: Comparison: Active Device vs Sham Device; Comparison for REM minutes. Group Selection refers to study device Condition (Active/Sham); repeated-measures design; Test type: Other — Effect size determination; Cohen's d = -0.82

2. Primary Outcome: Change in Sleep Architecture
Description: Percentage of each sleep stage defined by the American Academy of Sleep Medicine (NREM1, NREM2, NREM3, and REM), measured by clinically standard elements of Polysomnography and scored by a Registered Polysomnographic Technologist.
  Note: Randomization to Active or Sham during Phase 1 or Phase 2 occurred at the end of Baseline week.
Time Frame: The later viable night of two recordings: At the end of Phase 1 - Week 2 or Phase 1 - Week 3, and At the end of Phase 2 - Week 2 or Phase 2 - Week 3. Sleep stage percentage (relative to Latency to Persistent Sleep, Edinger et al. 2013).
Population: The same 10 (total) participants are represented in Arm/Group (repeated-measures)
Measure: Mean (Standard Deviation); unit: % of total sleep
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 10 | 10
% of total sleep
  NREM1 | 12.8 (6.7) | 13.0 (7.2)
  NREM2 | 55.5 (6.8) | 54.3 (9.5)
  NREM3 | 9.0 (7.4) | 5.9 (4.5)
  REM | 22.6 (6.3) | 26.8 (9.6)
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Comparison for NREM1 percentage. Group Selection refers to study device Condition (Active/Sham); repeated-measures design; Test type: Other — Effect size determination; Cohen's d = -0.04
Statistical Analysis 2: Comparison: Active Device vs Sham Device; Comparison for NREM2 percentage. Group Selection refers to study device Condition (Active/Sham); repeated-measures design; Test type: Other — Effect size determination; Cohen's d = 0.24
Statistical Analysis 3: Comparison: Active Device vs Sham Device; Comparison for NREM3 percentage. Group Selection refers to study device Condition (Active/Sham); repeated-measures design; Test type: Other — Effect size determination; Cohen's d = 0.80
Statistical Analysis 4: Comparison: Active Device vs Sham Device; Comparison for REM percentage. Group Selection refers to study device Condition (Active/Sham); repeated-measures design; Test type: Other — Effect size determination; Cohen's d = -0.78

3. Primary Outcome: Change in Insomnia Symptoms
Description: Self-reported score on the Insomnia Severity Index (ISI; 0-28) e-survey, where a higher score indicates worse/more Insomnia symptoms.
Time Frame: Sum ISI score near end of Phase 1 (study wks2-4) and near end of Phase 2 (study wks6-8).
Population: In this repeated-measures design, one participant had missing data for an Insomnia Severity Index (ISI) measure. Therefore, the analyzed sample for ISI Outcome is n=9 (5 Active Device Phase 1, then Sham; + 4 Sham Device Phase 1, then Active), rather than n=10.
Measure: Mean (Standard Deviation); unit: Sum score, on a scale of 0-28
Arm/Group | Active Device | Sham Device
Number analyzed (Participants) | 9 | 9
Sum score, on a scale of 0-28 | 7.3 (4.4) | 6.8 (5.0)
Statistical Analysis 1: Comparison: Active Device vs Sham Device; Group Selection refers to study device Condition (Active/Sham); repeated-measures design; Test type: Other — Effect size determination; Cohen's d = 0.11

ADVERSE EVENTS:
Time Frame: Systematic event monitoring occurred at a minimum of each scheduled polysomnography (night sleep monitoring) visit (6 total nights): twice during Baseline (1 week, at beginning and end), twice during Phase 1 (3 weeks, at end of 2nd week and end of 3rd week), and twice during Phase 2 (3 weeks, at end of 2nd week and at end of 3rd week). Non-systematic event monitoring also occurred throughout the 8 weeks of study data collection per participant, and across participants 9/28/2024 - 5/10/2024.
Description: The Adverse Event definition used in this research is the same as that used by clinicaltrials.gov. Adverse Event data were collected using a standard researcher-administered survey at study visits.
Arm/Group | Active Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Device (N=10) | Sham Device (N=10)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Bladder infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cornea tear (Eye disorders) | 0 (0) | 1 (1)
Aching, Discomfort, or Pain (various) (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Study watch discomfort (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stye (Eye disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment in this small pilot study was predominantly female (8/10), limiting the extension of effect size findings to a broader population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT05908344/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT05908344/ICF_002.pdf